CLINICAL TRIAL: NCT02102568
Title: Study of the Impact of Chemo-induced Menopause on the Quality of Life in Young Women of Childbearing Age and Diagnosed With Non-metastatic Breast Cancer
Brief Title: Impact of Chemo-induced Menopause on Quality of Life in Women <45 Years Old, Diagnosed With Non-metastatic Breast Cancer
Acronym: MENOCOR
Status: Completed | Type: Observational
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A01284-41
Record Dates: First submitted 2014-03-20; First posted 2014-04-03 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2021-08

CONDITIONS: BREAST CANCER
Keywords: breast cancer; Chemotherapy-induced menopause; quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum is collected in order to measure AMH (Anti-Müllerian Hormone) levels, before the start of chemotherapy and after the end of chemotherapy treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective multicenter study, Not on Health Products that evaluates up to 2 and a half years the impact of chemo-induced menopause (CIM) on the functional score of the QLQ-C30 quality of life questionnaire in young women of childbearing age, diagnosed with non-metastatic breast cancer.

DETAILED DESCRIPTION:
Approximately 20% of women with breast cancer are still of childbearing age and are likely to benefit from chemotherapy. Since Chemotherapy-Induced Menopause (CIM) may be one of its consequences, it seems important to study its impact on the quality of life of these young patients. It is within this framework that the Jean Perrin Center promoted the MENOCOR study, whose main objective is to assess the impact of the CIM on the quality of life through the QLQ-C30 functional score over a two-year period. The CIM incidence, its impact on quality of life (body image, anxiety, depression, physical activity and sleep quality) and the onset of climacteric signs, the onset of amenorrhea according to chemotherapy protocols and patient age and hormonal variations are among the secondary objectives of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 and under 45
* Patient without amenorrhea at diagnosis
* Performance status less than 2 (according to WHO criteria )
* Patient diagnosed with histologically proven non-metastatic breast cancer
* Clinical Stages I, IIA, IIB and IIIA
* Positive Hormone Receptors (defined by a rate of 10% of labeled cells and immunohistochemistry (IHC) ) or negative
* Positive or negative HER2 status ( defined a score of 0 or 1 + by IHC , or a 2 + score by IHC and FISH / ISHS / CISH negative)
* Patients to be treated with neoadjuvant or adjuvant chemotherapy
* Satisfying hematological, renal and hepatic functions : PNN> 2,109 / L, platelets > 100 . 109 / L, Hb> 10 g / dl , normal bilirubin, AST and ALT <2.5 upper normal value ( VNS) , alkaline phosphatase <2.5 VSN , creatinine clearance > 60 ml / min
* Obtaining informed consent in writing, signed and dated
* Affiliation to Social Security system (or being the beneficiary of such a plan) under the terms of the Act of August 9, 2004

Exclusion Criteria:

* Male patient
* Metastatic cancer
* Any T4 tumor (skin invasion, deep grip, inflammatory breast cancer)
* Patient who underwent surgical castration of ovariectomy or hysterectomy or tubal ligation
* Patients with endometriosis
* Pregnant or breastfeeding patients
* Patients with no effective contraception
* Patients who have had hormone therapy or chemotherapy
* Patient who have already taken Gn-RH or LH-RH analogues (chemical castration)
* Patient whose mother was in menopause early without treatment
* Presence of comorbidities related to fertility or medical history related to ovarian failure or sterility
* Significant neurological or psychiatric abnormalities
* Inability of the patient to complete the questionnaires (the language barrier)
* Patients deprived of liberty by court or administrative decision
* Patient with another pathology deemed incompatible with the inclusion of the patient in the protocol
* Participation in another clinical trial involving the chemical or surgical castration of the patient
* Patients geographically unstable in the 6 months following inclusion or residing away from the treatment center and thereby making it difficult to monitor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: premenopausal women with age between 18 to 45 years. premenopausal women with non-metastatic breast cancer.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2014-04; Primary Completion 2020-07-10 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the 2-year impact of chemo-induced menopause (CIM) on the functional score of the QLQ-C30 quality of life questionnaire in young women of childbearing age and diagnosed with breast cancer. | 3 years
  Differential variation of QLQ-C30 QoL Functional Score between inclusion and at 2 years.

SECONDARY OUTCOMES:
Evaluation of the rate of CIM after chemotherapy | 3 years
  Number of postmenopausal women after chemotherapy
Sensitivity and Specificity of blood Anti-Mullerian Hormone (AMH) in the prediction of MCI | 3 years
  Blood testing of AMH at baseline and post-chemotherapy
Predictive value of 6-month amenorrhea on 2-year menopause | 3 years
  Rate of patients recovering after 6 months of amenorrhea
Assessment of FSH (follicle stimulating hormone) and estradiol levels before chemotherapy and at the end of chemotherapy | 6 months
  Blood levels of FSH and estradiol at baseline and post-treatment
Impact of CIM on specific aspects of quality of life (anxiety, depression, body image, physical activity and quality of sleep) after breast cancer | 3 years
  Dimensional scores and overall scores of QLQ-BR23 (EORTC), HAD, BIQ (Body Image Questionnaire) questionnaires, Leeds sleep questionnaire, Ricci and Gagnon physical activity questionnaire
Time of onset of amenorrhea in terms of type of chemotherapy | 6 months to 1 year
  Time of onset of amenorrhea according to the type of chemotherapy (Kaplan-Meier method)
Time of onset of amenorrhea in terms of patient age | 6 months to 1 year
  Occurrence of MCI according to age
Differential variation of the symptomatic score of the QLQ-C30 questionnaire at 2 years according to menopausal status | 3 years
  QLQ-C30 Quality of Life Questionnaire Score
Longitudinal study of the quality of life of patients after treatment according to whether patients are menopausal or not | 3 years
  90/5000 Overall score of quality of life of patients at inclusion, at 1, 2 and 3 years post-inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Ange MOURET-REYNIER, Dr, Principal Investigator — Centre Jean Perrin
Locations (3):
- France (3):
  - Centre de lutte contre le cancer - Centre Jean PERRIN, Clermont-Ferrand
  - Institut Jean Godinot, Reims
  - CHU Saint Etienne, Saint-Etienne